CLINICAL TRIAL: NCT00940901
Title: Sildenafil for Treatment of Priapism in Men With Sickle Cell Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NA_00017554; RFA-HL-06-008 (Other Grant/Funding Number: Interdisciplinary Research Consortium U54)
Record Dates: First submitted 2009-07-16; First posted 2009-07-17 (Estimated); Results first posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Sickle Cell Disease; Priapism
Keywords: priapism; sickle cell disease; sildenafil; phosphodiesterase type 5 inhibitor
MeSH Terms: conditions — Anemia, Sickle Cell; Priapism | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sildenafil (Experimental): Participants assigned to this arm were given sildenafil 50 mg tablet daily for 16 weeks.
  Interventions: Drug: sildenafil
- placebo (Placebo Comparator): Participants assigned to this arm were given a placebo pill for the first 8 weeks, and then Sildenafil 50 mg for weeks 9-16.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: sildenafil — sildenafil 50 mg tablet daily for first 8 weeks (phase 1), and then sildenafil 50 mg tablet daily for final 8 weeks (phase 2)
  Other Names: Viagra
  Arms: sildenafil
Other: placebo — placebo 50 mg tablets daily for first 8 weeks (phase 1), and then sildenafil 50mg tablet daily for final 8 weeks (phase 2)
  Arms: placebo

SUMMARY:
This research is being done to evaluate if the phosphodiesterase type 5 (PDE5) inhibitor sildenafil has an effect on the frequency of recurrent priapism and the quality of life of males with sickle cell disease (SCD).

DETAILED DESCRIPTION:
The proposed research is designed to investigate the utility of continuous, long-term PDE 5 inhibitor therapy as an intervention for recurrent ischemic priapism, a disorder of non-willful, excessive penile erection, in patients with SCD. Although precise prevalence figures are not available, priapism in SCD is highly prevalent and thought to afflict approximately 40% of males, based on available literature. Additionally, the disorder exacts devastating consequences, including erectile tissue necrosis, erectile dysfunction, and psychological distress. Management of this disorder remains challenging because the mechanisms underlying priapism are incompletely understood.

ELIGIBILITY:
Inclusion Criteria:

* Ages 14 to 45, inclusive
* Episodes of prolonged penile erection in the absence of sexual interest or desire, with an average frequency of at least twice weekly, when averaged over the previous four weeks
* Able to provide informed consent or assent

Exclusion Criteria:

* Use of chronic nitrates or recreational use of nitrate containing products
* Use of a PDE5 (phosphodiesterase type 5)inhibitor within the previous two weeks
* Alcohol use exceeding two standard drinks daily
* Hypersensitivity to sildenafil
* Estimated glomerular filtration rate <50ml/min
* Known cirrhosis
* Retinitis pigmentosa
* Necessary use of a P450 3A4 inhibitor (a drug which can increase plasma levels of sildenafil when taken together)

Ages: 14 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2008-06; Primary Completion 2012-11 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur L. Burnett, MD, MBA, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Then Sildenafil: Participants assigned to this arm were given a placebo pill for the first 8 weeks, and then Sildenafil 50 mg for weeks 9-16.
Period: Weeks 1-8 (Phase 1)
Arm/Group | Sildenafil | Placebo Then Sildenafil
Started | 6 | 7
Completed | 6 | 7
Not Completed | 0 | 0
Period: Week 9-16 (Phase 2)
Arm/Group | Sildenafil | Placebo Then Sildenafil
Started | 6 | 7
Completed | 4 | 4
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sildenafil | Placebo Then Sildenafil | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.7 (5.3) | 23.0 (8.7) | 22.5 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 7 | 13
Region of Enrollment [Number; unit: participants]
  United States | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Greater Than or Equal to a 50% Reduction in Priapic Episodes
Description: A "Priapism sexual activity log" was administered to participants. In the log, participants were asked to quantify the number of priapic episodes they had experienced in the previous 2 weeks according to the following scale/tiers: 0 = no episodes, 1 = 1-2 episodes, 2 = 3-4 episodes, 3 = 5-8 episodes and 6 = greater than 20 episodes.
Time Frame: change between baseline and 8 weeks post intervention
Population: Intention to treat analysis.
Measure: Number; unit: Number of participants
Arm/Group | Sildenafil | Placebo Then Sildenafil
Number analyzed (Participants) | 6 | 7
Number of participants | 3 | 3
Statistical Analysis 1: Comparison: Sildenafil vs Placebo Then Sildenafil; Null hypothesis: there would be no difference in the number of participants who experienced at least a 50% reduction in the frequency of priapic episodes between baseline and 8 weeks post intervention, between the sildenafil and placebo groups; Test type: Superiority or Other; p = 1, Fisher Exact

2. Primary Outcome: Greater Than or Equal to a 50% Reduction in Priapic Episodes
Description: as for outcome 1
Time Frame: change between 8 weeks post intervention and 16 weeks post intervention
Population: 3 participants from the Phase 1 Sildenafil group were lost to follow up during the second phase; 2 individuals from the Phase 1 Placebo then sildenafil group were lost to follow up during the second phase.
Measure: Number; unit: Number of participants
Arm/Group | Sildenafil | Placebo Then Sildenafil
Number analyzed (Participants) | 4 | 4
Number of participants | 2 | 3
Statistical Analysis 1: Comparison: Sildenafil vs Placebo Then Sildenafil; Test type: Superiority or Other; p = 0.55, Fisher Exact

ADVERSE EVENTS:
Time Frame: baseline to 16 weeks post intervention
Groups:
- Sildenafil Phase 1; Sildenafil Phase 2: Participants taking sildenafil 50 mg tablet daily for weeks 1-8 during Phase 1 and during weeks 9-16 during Phase 2
- Placebo Then Sildenafil Phase 1; Placebo Then Sildenafil Phase 2: Participants taking placebo daily for weeks 1-8 during phase 1 then taking Sildenafil 50mg tablet daily for weeks 9-16 during phase 2
Arm/Group | Sildenafil Phase 1 | Placebo Then Sildenafil Phase 1 | Sildenafil Phase 2 | Placebo Then Sildenafil Phase 2
Serious Adverse Events (participants affected / at risk) | 3/6 | 1/7 | 1/4 | 0/4
Other Adverse Events (participants affected / at risk) | 5/6 | 5/7 | 2/4 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sildenafil Phase 1 (N=6) | Placebo Then Sildenafil Phase 1 (N=7) | Sildenafil Phase 2 (N=4) | Placebo Then Sildenafil Phase 2 (N=4)
Priapism (Blood and lymphatic system disorders) | 2 (4) | 1 (1) | 1 (1) | 0 (0)
lightheadedness (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
shortness of breath (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
coffee ground emesis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
emesis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
epistaxis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
fever (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
chills (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
back pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
chest tightness (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
rhinorrhea (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
cough (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
congestion (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
asthma attack (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaso-occlusive Pain crisis (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Penile Swelling (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Low blood count (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sildenafil Phase 1 (N=6) | Placebo Then Sildenafil Phase 1 (N=7) | Sildenafil Phase 2 (N=4) | Placebo Then Sildenafil Phase 2 (N=4)
Priapism (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 2 (3) | 0 (0)
vision trouble (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
jittery feelings (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
viral upper respiratory infection/cough/sore throat (cold) (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2) | 1 (1) | 0
stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
low blood count (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
elevated temperature (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
pain crisis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No